CLINICAL TRIAL: NCT04467151
Title: A Randomized, Double-blind, Placebo-controlled Trial of Anti-SARS-CoV-2 Plasma in Hospitalized Non-ICU Patients With COVID-19
Brief Title: Administration of Anti-SARS-CoV-2 Convalescent Plasma in Hospitalized, Non-ICU Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not obtain funding to proceed with study
Sponsor: Kashif Khan (Other)
Responsible Party: Sponsor-Investigator, Kashif Khan, Principal Investigator, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-20-00516
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: Anti-SARS-CoV-2 plasma
MeSH Terms: conditions — COVID-19 | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- anti-SARS-CoV-2 plasma (Experimental): Patients receive one dose (250-300ml) of anti-SARS-CoV-2 convalescent plasma
  Interventions: Drug: anti-SARS-CoV-2 plasma
- Placebo (Placebo Comparator): Patients receive one dose (250-300ml) of placebo (albumin 5%)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: anti-SARS-CoV-2 plasma — Administration of anti-SARS-CoV-2 convalescent plasma
  Other Names: Convalescent Plasma
  Arms: anti-SARS-CoV-2 plasma
Other: Placebo — Administration of placebo (albumin 5%)
  Other Names: Albumin
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the administration of anti-SARS-CoV-2 convalescent plasma in COVID-19 patients who are sick enough to warrant hospitalization, but not yet admitted to the ICU (prior to the onset of overwhelming disease including a systemic inflammatory response, sepsis, and/or ARDS).

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of anti-SARS-CoV-2 convalescent plasma in COVID-19 patients.

After confirmation of COVID-19, patients that meet the eligibility requirement and provide informed consent will be randomized in a 2:1 ratio to anti-SARS-CoV-2 convalescent plasma (1 unit of approximately 250 ml) or placebo (1 unit albumin 5%, approximately 250 ml). We will evaluate the ability of anti-SARS-CoV-2 convalescent plasma vs. placebo control to decrease disease progression (measured by the WHO Ordinal Scale for Clinical Improvement) during the 28 days following administration to hospitalized, non-ICU patients. If patient is discharged from the hospital prior to Day 28, Day 28 assessment will be by phone.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Hospitalized with COVID-19-related acute respiratory symptoms
* Initial COVID-19 severity status on the WHO Ordinal Scale for Clinical Improvement = 3 ("Hospitalized, no oxygen therapy) or 4 ("Hospitalized, on oxygen by mask or nasal prongs")
* Laboratory-confirmed COVID-19
* First signs of infection occurring no more than 14 days prior to enrollment

Exclusion Criteria:

* Receipt of pooled immunoglobulin in the past 30 days
* Contraindication to transfusion or history of prior reactions to transfusion blood products
* Admission to intensive care unit at any point during hospital course prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression measured by WHO scale | Day 0 through Day 28 (or hospital discharge)
  Disease progression from the state at randomization (with a "3" or "4" on the WHO Ordinal Scale for Clinical Improvement) to requiring invasive mechanical ventilation (which is "6" or greater on the WHO scale) during the study period

SECONDARY OUTCOMES:
Comparison of maximum WHO score per group | Day 0 through Day 28 (or hospital discharge)
  Comparison of the number of participants reaching a maximum daily WHO score of 5, 7, and 8 during the study period per group
Comparison of decrease of median and maximum WHO score per group | Day 0 through Day 28 (or hospital discharge)
  Comparison of the median and maximum daily WHO scores during the study period per group
Comparison of time to clinical improvement per group | Day 0 through Day 28 (or hospital discharge)
  Comparison of time to clinical improvement, defined as time between randomization and time to improvement (WHO Ordinal Scale "2" first reached for at least 1 day)
Comparison of time to reach score of "6" or greater on the WHO scale | Day 0 through Day 28 (or hospital discharge)
  Evaluate the time to reach score of at least 6 within 28 days

OTHER OUTCOMES:
Comparison of hospital length of stay per group | Day 0 through Day 28 (or hospital discharge)
  Evaluate number of days hospitalized
Comparison of ICU length of stay per group | Day 0 through Day 28 (or hospital discharge)
  Evaluate number of hours in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Kashif T Khan, MD, SM, Principal Investigator — Keck School of Medicine of University of Southern California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Casadevall A, Pirofski LA. The damage-response framework of microbial pathogenesis. Nat Rev Microbiol. 2003 Oct;1(1):17-24. doi: 10.1038/nrmicro732. PMID 15040176
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] van Griensven J, Edwards T, Gallian P; Ebola-Tx Consortium. Convalescent Plasma for Ebola Virus Disease. N Engl J Med. 2016 Jun 23;374(25):2500. doi: 10.1056/NEJMc1602284. No abstract available. PMID 27332913
- [Background] Zhang B, Liu S, Tan T, Huang W, Dong Y, Chen L, Chen Q, Zhang L, Zhong Q, Zhang X, Zou Y, Zhang S. Treatment With Convalescent Plasma for Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Chest. 2020 Jul;158(1):e9-e13. doi: 10.1016/j.chest.2020.03.039. Epub 2020 Mar 31. PMID 32243945